CLINICAL TRIAL: NCT03874442
Title: The Effectiveness of a Preoperative, Interactive Game: "SERES Pain in Children" to Decrease the Perioperative Pain and Anxiety Level in Children
Brief Title: The Effectiveness of a Preoperative, Interactive Game "SERES Pain in Children".
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, karel allegaert, Prof. Dr. Neonatology, Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: S58541
Record Dates: First submitted 2019-03-08; First posted 2019-03-14 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Ambulatory Surgery in Children
Keywords: postoperative pain in children; preoperative anxiety in children

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Controls (No Intervention)
- CliniPup (Experimental)
  Interventions: Other: CliniPup serious game

INTERVENTIONS:
Other: CliniPup serious game — The interactive game is played at home by the children on a computer or tablet before the surgery. The "SERES Pain in Children"-game is created with realistic scenarios based on scientific literature about perioperative pain and fear in children. The primary goal of the game is to provide the children insight in the impact of their personal choices on their well-being and on their environment by giving the children information about the day of the surgery. The ultimate aim of the game is to create a change in behaviour, enhance children's coping strategies and reduce the burden of pain and fear in the children and parents.
  Arms: CliniPup

SUMMARY:
Perioperative pain and fear in children is an important health problem in our society, both at the time of surgery and in their future life. Nonetheless, the management of perioperative pain and fear in children is still challenging and poorly addressed.

Bad management of perioperative pain and fear can lead to traumatic events. This might result in an increased morbidity and mortality on the long term, as these patients do wait significantly longer than control subjects to consult medical services (1).

Previous evidence has shown that preoperative fear, in both children and parents, is a significant determinant of perioperative pain (2). Other studies revealed that pain and fear are strongly related; higher preoperative stress can result in higher postoperative pain scores (3).

This shows the need for a constructive, effective and clear tool to guide children through their perioperative experience. Mindbytes created a serious game, "SERES Pain in Children", to address this need.

Serious gaming is a way of learning, training and educating using gaming principles. Young persons, growing up around computers, are especially eligible for gaming. Therefore serious gaming is a strategy to catch their attention and educate them in a playful manner. Serious gaming is even incorporated in higher education and corporate entities. There are also a few examples of serious games for training healthcare providers, supporting patients in their therapy, disease management or even to promote healthy wellness and lifestyle to the broader public (4,5).

The "SERES Pain in Children"-game is created with realistic scenarios based on scientific literature about perioperative pain and fear in children. The primary goal of the game is to provide the children insight in the impact of their personal choices on their well-being and on their environment by giving the children information about the day of the surgery. The ultimate aim of the game is to create a change in behaviour, enhance children's coping strategies and reduce the burden of pain and fear in the children and parents.

The overall objective of this study is to investigate the effectiveness of the implementation of an interactive preparative 'serious' game to decrease the perioperative distress in children. Our aim is to validate this game by investigating the level of discomfort in children and care providers who played the game before surgery compared to control subjects who did not play the game.

DETAILED DESCRIPTION:
Background Perioperative pain and fear in children is an important health problem in our society, both at the time of surgery and in their future life. Nonetheless, the management of perioperative pain and fear in children is still challenging and poorly addressed.

Bad management of perioperative pain and fear can lead to traumatic events. This might result in an increased morbidity and mortality on the long term, as these patients do wait significantly longer than control subjects to consult medical services (1).

Previous evidence has shown that preoperative fear, in both children and parents, is a significant determinant of perioperative pain (2). Other studies revealed that pain and fear are strongly related; higher preoperative stress can result in higher postoperative pain scores (3).

This shows the need for a constructive, effective and clear tool to guide children through their perioperative experience. Mindbytes created a serious game, "SERES Pain in Children", to address this need.

Serious gaming is a way of learning, training and educating using gaming principles. Young persons, growing up around computers, are especially eligible for gaming. Therefore serious gaming is a strategy to catch their attention and educate them in a playful manner. Serious gaming is even incorporated in higher education and corporate entities. There are also a few examples of serious games for training healthcare providers, supporting patients in their therapy, disease management or even to promote healthy wellness and lifestyle to the broader public (4,5).

The "SERES Pain in Children"-game is created with realistic scenarios based on scientific literature about perioperative pain and fear in children. The primary goal of the game is to provide the children insight in the impact of their personal choices on their well-being and on their environment by giving the children information about the day of the surgery. The ultimate aim of the game is to create a change in behaviour, enhance children's coping strategies and reduce the burden of pain and fear in the children and parents.

Main objective The overall objective of this study is to investigate the effectiveness of the implementation of an interactive preparative 'serious' game to decrease the perioperative distress in children. Our aim is to validate this game by investigating the level of discomfort in children and care providers who played the game before surgery compared to control subjects who did not play the game.

ELIGIBILITY:
Inclusion Criteria:

* Male/female
* Age: 6 - 10 years
* Parents have to sign an informed consent
* Children have to give their assent
* Children and parents have to understand and speak Dutch

Exclusion Criteria:

* Children who suffer from a mental illness
* Children who have a developmental delay
* Children who have a history of affective disorder
* Children with an ASA (American Society of Anesthesiology) physical status higher than II

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2016-02-22 (Actual); Primary Completion 2016-04-26 (Actual); Study Completion 2016-04-26 (Actual)

PRIMARY OUTCOMES:
Preoperative anxiety | at the hospital before surgery
  Perioperative anxiety measured with the mYPAS
Postoperative pain | after surgery
  Children were asked to scale their pain using the WBFPRS once they were awake and responsive (15 minutes after they were back in their room). The WBFPRS is used to assess pain in children and help them communicate about it [26]. The WBFPRS, which is an auto-evaluation scale, has six faces representing "no pain" (0) to "worst pain ever".

SECONDARY OUTCOMES:
User experience and satisfaction | At the hospital, before surgery
  user experience and satisfaction was also assessed through a questionnaire wherein parents and children completed a Likert scale for each question. Additionally, parents were asked to which extent they would recommend CliniPup to peers and a net-promoter score (NPS) was calculated.
parental anxiety | At the hospital, before surgery
  After signing the consent and assent papers, parental anxiety was assessed with the STAI, a widely used self-report anxiety-assessment instrument.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Buffel C, van Aalst J, Bangels AM, Toelen J, Allegaert K, Verschueren S, Vander Stichele G. A Web-Based Serious Game for Health to Reduce Perioperative Anxiety and Pain in Children (CliniPup): Pilot Randomized Controlled Trial. JMIR Serious Games. 2019 Jun 1;7(2):e12431. doi: 10.2196/12431. PMID 31199324